CLINICAL TRIAL: NCT00032968
Title: Buprenorphine/Naloxone Versus Clonidine For Out-patient Opiate Detoxification
Brief Title: Buprenorphine/Naloxone Versus Clonidine for Outpatient Opiate Detoxification - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Walter Ling, M.D., University of California, Los Angeles
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0002-1; NCT00016757 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Heroin Dependence; Morphine Dependence; Substance Withdrawal Syndrome
Keywords: opiate dependence
MeSH Terms: conditions — Heroin Dependence; Morphine Dependence; Substance Withdrawal Syndrome; Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to assess buprenorphine/naloxone versus clonidine for outpatient opiate detoxification.

DETAILED DESCRIPTION:
Patients randomized to the BUP/NX arm will receive daily doses for 13 days with sublingual administration of 2 mg buprenorphine/0.5 mg naloxone tablet(s) and/or an 8 mg buprenorphine/2.0 mg naloxone tablet(s). The starting dose on day 1 is 4 mg/1 mg BUP/NX with an additional 4 mg/1 mg, if needed, escalating in a step-wise manner to 16 mg/4 mg BUP/NX on day 3 and tapering to 2 mg/ 0.5 mg BUP/NX by days 12 to 13. Patients randomized to the clonidine arm will receive oral clonidine (0.05 to 0.1 mg depending upon weight) every 4 to 6 hours for 24 hours not to exceed 0.6 mg total on day 1. On day 2, a clonidine transdermal patch will be applied (0.1 mg/day/7-day patch with number of patches adjusted by weight). Oral clonidine will continue to be given on the second day of detoxification and increased to 0.2 mg every 6 hours or 0.1 mg every 3 hours not to exceed 0.8 mg over 24 hours. Patches will be worn all 13 days of detoxification. The dose of clonidine will be adjusted according to the proposed detoxification schedule, patient's weight, tolerance, and systolic blood pressure. Patients will receive counseling according to procedures in existence at each CTP throughout the study. Self-help detoxification handbooks will be distributed to all study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-seeking males and non-pregnant and non-lactating females, 15 years and older, who fulfill DSM-IV criteria for opiate dependence, report experiencing symptoms of opiate withdrawal, are currently physically dependent on opioids and are in need of medical assistance for opioid withdrawal.
2. Systolic blood pressure 100 mm Hg, and pulse 56 bpm.
3. Good general health or, in case of a medical/psychiatric condition needing ongoing treatment, under the care of a physician willing to continue patient's medical management and cooperate with the study physicians.
4. Agreeable to and capable of signing the informed consent approved by an institutional review board and, if under the age of 18 (excluding emancipated minors), assent and concurrent consent from a parent or legal guardian.
5. Use of one of the following acceptable methods of birth control by female patients of childbearing potential:

   1. oral contraceptives
   2. barrier (diaphragm or cervical cap) with spermicide or condom
   3. intrauterine progesterone contraceptive system
   4. levonorgestrel implant
   5. medroxyprogesterone acetate contraceptive injection
   6. complete abstinence from sexual intercourse

Exclusion Criteria:

1. Medical condition that would make participation, in the opinion of the study physician, medically hazardous (e.g., acute hepatitis, unstable cardiovascular, liver or renal disease);
2. Clinically significant abnormalities in ECG.
3. Known allergy or sensitivity to buprenorphine, naloxone, or clonidine.
4. Receiving beta-blockers, calcium channel blockers, tricyclics, digitalis and other medications which may interact adversely with clonidine.
5. Acute severe psychiatric condition in need of immediate treatment, or imminent suicide risk.
6. Dependence on alcohol, benzodiazepines or other depressants, or stimulants, and requiring immediate medical attention.
7. Participation in an investigational drug study, including buprenorphine, within the past 30 days.
8. Methadone or LAAM maintenance or detoxification within 30 days of enrollment.
9. Pending legal action that could prohibit or interfere with participation.
10. Unable to remain in area for duration of active phase of treatment.
11. Females that are pregnant, lactating, or planning to become pregnant.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341
Dates: Start 2001-01; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Degree of drug craving
Opiate craving
Adverse events
Drug craving
Decreased frequency of HIV related behavior
Adverse effect measures

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Los Angeles Treatment Research Center
Locations (7):
- United States (7):
  - Haight-Ashbury Free Clinic, Berkeley, California
  - Aegis Medical Systems, Inc., Oxnard, California
  - Midtown Community Mental Health Center, Indianapolis, Indiana
  - UMDNJ - Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Bellevue, New York, New York
  - Kaiser Permanente Northwest, Division of Addiction, Portland, Oregon

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0002